CLINICAL TRIAL: NCT02924285
Title: CAT-PVC Trial Catheter Ablation Versus Amiodarone for Therapy of Premature Ventricular Contractions in Patients With Structural Heart Disease: a Randomized Trial
Brief Title: Catheter Ablation Versus Amiodarone for Therapy of Premature Ventricular Contractions in Patients With Structural Heart Disease
Acronym: CAT-PVC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Helios Health Institute GmbH (Other); Abbott Medical Devices (Industry); Zentrum für Klinische Studien Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAT-PVC01
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Heart Diseases; Cardiomyopathies; Ventricular Premature Complexes
MeSH Terms: conditions — Heart Diseases; Cardiomyopathies; Ventricular Premature Complexes | interventions — Catheter Ablation; Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Procedure (Active Comparator): Radiofrequency catheter ablation
  Interventions: Procedure: Procedure (Radiofrequency catheter ablation)
- Antiarrhythmic Drug (Active Comparator): Amiodarone
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Procedure: Procedure (Radiofrequency catheter ablation) — Radiofrequency catheter ablation
  Arms: Procedure
Drug: Amiodarone — Amiodarone, Verification of superiority of catheter ablation over amiodarone for treatment of PVCs in patients with structural heart disease as:
  Antiarrhythmic Drug Amiodarone
  Arms: Antiarrhythmic Drug

SUMMARY:
For therapy of symptomatic premature ventricular complexes (PVCs) in subjects with structural heart disease the current European Guidelines for the management of patients with ventricular arrhythmias and the prevention of second cardiac death recommend catheter ablation as well as amiodarone with a class IIa indication. Due to the lack of randomized data this study investigates the comparison of catheter ablation and amiodarone for PVC treatment in patients with structural heart disease. Therefore, patients will be randomized to one of two treatment strategies: 1) catheter ablation, or 2) amiodarone.

DETAILED DESCRIPTION:
Premature ventricular contractions (PVCs) are frequently encountered in patients with or without structural heart disease. Even though PVCs in healthy subjects are considered to be a benign arrhythmia. There is also evidence for the risk of a reversible cardiomyopathy due to the PVC-induced inter- and intraventricular dyssynchrony. Data show that elimination of PVCs by catheter ablation leads to an improvement of left ventricular dysfunction. In one-half of the heart failure patients frequent PVCs occur with more than 1000/24 h. In patients with structural heart disease premature ventricular contractions (PVCs) lead to an increased mortality risk with only a burden of 10 PVC per hour. Further decreasing of left ventricular function and worsening of heart failure are described. Therefore, therapy of frequent monomorphic PVCs is recommended in these subjects. Beta-blockers as part of standard therapy often remain ineffective or may lead to a paradoxic effect in patients with bradycardia. A limiting factor for selection of antiarrhythmic drug due to increasing mortality is the presence of structural heart disease. So in the most cases amiodarone is indicated. There are data showing improvement of LV function after suppression of PVCs by amiodarone with a significant reduction of the PVC burden in comparison to baseline. However, the adverse effects of amiodarone are well-known especially in long-term therapy. On the other hand, radiofrequency catheter ablation is a widely applied and safe treatment option for PVCs with a high acute success rate of up to 90% PVC reduction in various circumstances like pre-existing heart failure and post myocardial infarction subjects. Some small-sample studies show the benefit of catheter ablation in subjects with depressed LV function. To date, there are no randomized data for comparison of catheter ablation and amiodarone for therapy of PVCs in patients with structural heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Structural heart disease with or without left ventricular dysfunction with
* PVCs on Holter monitoring (burden >10.000/d) AND/OR
* PVCs on Holter monitoring correlating with symptoms AND/OR
* Reduction of biventricular pacing <92% in subjects with implanted cardiac resynchronization therapy (CRT) device
* Age: 18-87 years
* Willing and capable of giving informed consent

Exclusion Criteria:

* Previous ablation procedure or amiodarone for PVC without success
* New York Heart Association (NYHA) functional class IV
* Intracardial thrombus
* Pulmonary fibrosis
* Liver cirrhosis ≥ CHILD B
* Manifest hyper- or hypothyreoidism
* Long QT (QTc > 500 ms if QRS<120 ms, if QRS>120 ms according to QTRR, QRS formula)
* Sick sinus syndrome with symptomatic bradycardia <55 bpm or AV node conduction delay without implanted pacing device
* Known side effects under amiodarone or iodine
* Idiopathic angioedema
* Comedication with known risk for torsade-de-pointes tachycardia
* Pregnancy or lactation

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Verification of superiority of catheter ablation over amiodarone for treatment of PVCs in patients with structural heart disease | Baseline and after 6 weeks
  difference of the PVC burden in a 24 h Holter registration after 6 weeks and at baseline expressed as the amount of the baseline value ΔVES_r = (VES_6 - VES_0) / VES_0

SECONDARY OUTCOMES:
Change in quality of life (QoL) score according EQ-5D questionnaire | Baseline, after 6 weeks and 12 months
Change in 6 minute walking distance | Baseline, after 6 weeks and 12 months
Change in left ventricular ejection fraction (LVEF) | Baseline, after 6 weeks and 12 months
Change in serum NT-proBNP level | Baseline, after 6 weeks and 12 months
Change in New York Heart Association (NYHA) functional class | Baseline, after 6 weeks and 12 months
Occurrence of cardiovascular related hospitalization | after 6 weeks and 12 months
Occurrence of drug adverse effects | after 6 weeks and 12 months
Occurrence of procedure related complications | after 6 weeks and 12 months
Difference of the PVC burden in a 24 h Holter registration after 12 months and at baseline expressed as the amount of the baseline value | Baseline and after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, MD, Principal Investigator — Heart Center Leipzig
Locations (1):
- Heart Center Leipzig, Leipzig, Germany